CLINICAL TRIAL: NCT02644681
Title: Neurophysiological Intraoperative Monitoring During Aortic Surgery
Acronym: NIMAS
Status: Completed | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Chiesa Roberto, Professor, Scientific Institute San Raffaele
Other Study IDs: NIMAS/32/OSR
Record Dates: First submitted 2015-12-04; First posted 2016-01-01 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic | interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Aortic Aneurysm, Thoracic surgery

SUMMARY:
The primary objective of this study is to evaluate if the motor-evoked potentials/motor action potential amplitude ratio and motor action potential amplitude measurement are useful in detecting spinal cord ischemia during thoracoabdominal aortic aneurysms surgery.

The secondary objective is to evaluate the presence of a correlation between neurophysiological changes and other factors (such as surgical maneuvers, anesthetic and physiologic changes) in order to find which factor is the most important in determining spinal cord ischemia.

This study is an observational, single-center, prospective study on patients with thoracoabdominal aortic aneurysms undergoing surgical repair with intraoperative motor-evoked potentials and somatosensory evoked potentials monitoring.

ELIGIBILITY:
Inclusion Criteria:

* satisfied criteria for Intraoperative neurophysiological monitoring;
* sign a written informed consent to participate in the study.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all consecutive patients with thoracoabdominal aortic aneurysms who will be subjected to neuromonitoring-guided open repair of the aortic aneurysm at the Department of Vascular Surgery of San Raffaele Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the motor-evoked potentials/motor action potential amplitude ratio | During thoracoabdominal aortic aneurysms surgery
  The goal of this study is to evaluate the efficacy of different neurophysiological parameters in predicting patient outcome. In particular, our objective is to verify if a better identification of peripheral nerve ischemia during TAAA procedure can improve the sensibility of Intraoperative neurophysiological monitoring in detecting spinal cord ischemia and predicting clinical outcome.
  Exploratory univariate analyses will be performed using logistic regression to calculate odds ratios to evaluate neurophysiological parameters associated with poor outcome. Factors that will be found to be significant at p < 0.05 will be then examined in subsequent multivariate analyses to determine significant independent predictors of poor outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy